CLINICAL TRIAL: NCT06125639
Title: Effects of Sauna Bathing on Sleep, Mood and Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWF_SKN_1
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sauna Group (Experimental)
  Interventions: Behavioral: Sauna Bathing
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Sauna Bathing — Participants will take part in 9 evening sauna bathing session over the course of 3 weeks
  Arms: Sauna Group

SUMMARY:
Sauna bathing is a popular, low-cost, and easily accessible type of whole-body thermotherapy that has been used for social, religious, health, and hygienic reasons for thousands of years. There is strong evidence to support the various physiological and psychological benefits of sauna bathing. The positive effects of regular sauna use have been explained by a number of mechanisms of action, including increased cardiac output, reduced peripheral vascular resistance and other physiological changes in cardiovascular parameters such as decreased systolic and/or diastolic blood pressure. Additionally, the psychological impact of sauna bathing may occur due to a combination of factors that include the release of endorphins, relaxation, placebo effects, and psychological and social interactions that likely occur around frequent sauna activity. Taken together, it is possible that acute and regular sauna bathing may impact sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* good general health assessed by physician
* written consent to participate

Exclusion Criteria:

* medication or dietary supplements, which could potentially impact the study outcomes
* history of sleep or neurological disorders
* regular sauna use
* professional athlete
* shift worker

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Objective Sleep - Time in bed | 5 weeks
  Total time spent in bed during the night assessed by sleep radar
Objective Sleep - Sleep-onset latency | 5 weeks
  The time it takes from when the participant intends to go to sleep and actually starts to sleep assessed by sleep radar
Objective Sleep - Total sleep time | 5 weeks
  Total sleep time obtained from sleep onset to time at wake-up assessed by sleep radar
Objective Sleep - Light sleep | 5 weeks
  Total amount of time in light sleep assessed by sleep radar
Objective Sleep - Deep sleep | 5 weeks
  Total amount of time in deep sleep assessed by sleep radar
Objective Sleep - REM sleep | 5 weeks
  Total amount of time in REM sleep assessed by sleep radar
Objective Sleep - Sleep efficiency | 5 weeks
  The percentage of total sleep time to lights off and leaving bed assessed by sleep radar

SECONDARY OUTCOMES:
Subjective Sleep Quality assessed by Karolinska Sleep Diary | 5 weeks
Stress level assessed by VAS scale | 5 weeks
  VAS scale is a 11-item self-report measure for stress. Answers range from 0 (no stress) to 10 (worst stress).
Positive and Negative Affect Schedule (PANAS) | baseline, after 1,3,6,9 sauna bathing, after 5 weeks
  The PANAS is a 20-item self-report measure for positive and negative affect.
Mood | baseline, after 1,3,6,9 sauna bathing, after 5 weeks
  Mood Adjective Check List (UMACL) will be used to assess mood (Mathews, Chamberlain & Jones, 1990, adapted to Polish by Ewa Goryńska, 2005). UMACL measures mood in three dimensions of the core affect: Tense Arousal (minimum value: 9, maximum value: 36), Energetic Arousal (minimum value: 10, maximum value: 40), and Hedonic Tone (minimum value: 10, maximum value: 40), with higher scores representing higher levels of the mood dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- University School of Physical Education in Cracow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No